CLINICAL TRIAL: NCT07076160
Title: Pilot Dispensing Study of Two Marketed Daily Disposable Multifocal Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-6612
Record Dates: First submitted 2025-07-14; First posted 2025-07-22 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Visual Acuity; Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Test/Control/Control (Experimental): Eligible subjects will be randomized into the Test/Control/Control sequence.
  Interventions: Device: INFUSE® One Day Multifocal; Device: ACUVUE® OASYS MAX 1-Day Multifocal Contact Lens
- Control/Test/Test (Experimental): Eligible subjects will be randomized into the Control/Test/Test sequence.
  Interventions: Device: INFUSE® One Day Multifocal; Device: ACUVUE® OASYS MAX 1-Day Multifocal Contact Lens

INTERVENTIONS:
Device: INFUSE® One Day Multifocal — Test Lens
Device: ACUVUE® OASYS MAX 1-Day Multifocal Contact Lens — Control Lens

SUMMARY:
This is a 6-visit, single-masked, multi-site, 2×3 crossover, randomized-controlled, dispensing clinical trial to evaluate visual acuity.

ELIGIBILITY:
Potential subjects must satisfy all of the following criteria to be enrolled in the study:

1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. Be at least 40 years of age and not greater than 70 years of age at the time of consent.
4. Own a wearable pair of spectacles if required for their distance vision.
5. Be an adapted soft contact lens wearer in both eyes (i.e. worn lenses a minimum of 2 days per week for at least 6 hours per wear day, for 30 days or more duration).
6. Either already be wearing a presbyopic contact lens correction (e.g., reading spectacles over contact lenses, monovision or multifocal contact lenses, etc.) or if not respond positively to at least one symptom on the "Presbyopic Symptoms Questionnaire".
7. The subject's distance spherical equivalent refraction must be in the range of +1.00 to +4.00 or -1.00 D to -4.00 D in each eye.
8. The subject's refractive cylinder must be ≤0.75 D in each eye.
9. The subject's ADD power must be in the range of +0.75 D to +2.50 D.
10. The subject must have distance best corrected visual acuity of 20/20-3 or better in each eye.

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

1. Be currently pregnant or lactating.
2. Have any active or ongoing ocular or systemic allergies that may interfere with contact lens wear.
3. Have been diagnosed with diabetes.
4. Have any active or ongoing systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear. This includes, but not be limited to, hyperthyroidism, Sjögren's syndrome, xerophthalmia, acne rosacea, Stevens-Johnson syndrome, and immunosuppressive diseases or any infectious diseases (e.g. hepatitis, tuberculosis).
5. Have any previous, or planned, ocular or intraocular surgery (e.g. radial keratotomy, PRK, LASIK, lid procedures, dacryocystorhinostomy, peripheral iridotomy/iridectomy, cataract surgery, retinal surgery, etc.).
6. Have a history of amblyopia, strabismus or binocular vision abnormality.
7. Use of any of the following medications within 1 week prior to enrollment: oral retinoid, oral tetracyclines, anticholinergics, oral phenothiazines, oral/inhaled corticosteroids. See section 9.1 for further examples.
8. Be currently using any ocular medications with the exception of rewetting drops.
9. Have a history of herpetic keratitis.
10. Have a history of irregular cornea.
11. Have a history of pathological dry eye.
12. Have participated in any contact lens or lens care product clinical trial within 7 days prior to study enrollment.
13. Be an employee (e.g., Investigator, Coordinator, Technician) or immediate family member of an employee (including partner, child, parent, grandparent, grandchild, sibling of the employee or their spouse) of the clinical site.
14. Have any known hypersensitivity or allergic reaction to non-preserved rewetting drop solutions or sodium fluorescein.
15. Have clinically significant (grade 3 or higher on the FDA grading scale) slit lamp findings (e.g., corneal edema, neovascularization or staining, tarsal abnormalities or bulbar injection) or other corneal or ocular disease or abnormalities that contraindicate contact lens wear or may otherwise compromise study endpoints (including entropion, ectropion, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, moderate or above corneal distortion, herpetic keratitis).
16. Have any current ocular infection or inflammation.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2025-07-24 (Actual); Primary Completion 2025-09-20 (Actual); Study Completion 2025-09-20 (Actual)

PRIMARY OUTCOMES:
High Luminance, High Contrast (HLHC) Binocular logMAR Visual Acuity at distance (4 meters) | 1-week follow-up
  Visual acuity after approximately 1-week in the optimized lens pair under HLHC illuminance conditions will be evaluated at distance (4 meters) using ETDRS Charts.
High Luminance, High Contrast (HLHC) Binocular logMAR Visual Acuity at intermediate (64 cm) | 1-week follow-up
  Visual acuity after approximately 1-week in the optimized lens pair under HLHC illuminance conditions will be evaluated at intermediate (64 cm) using reduced Guillon-Poling charts.
High Luminance, High Contrast (HLHC) Binocular logMAR Visual Acuity at near (40 cm) | 1-week follow-up
  Visual acuity after approximately 1-week in the optimized lens pair under HLHC illuminance conditions will be evaluated at near (40 cm) using reduced Guillon-Poling charts.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (7):
- United States (7):
  - Dr. James Weber & Associates, PA - City Square Blvd, Jacksonville, Florida
  - VRC, Jacksonville, Florida
  - Pearson Research Center, PA, Longwood, Florida
  - Maitland Vision Center - North Orlando Ave, Maitland, Florida
  - Sacco Eye Group, Vestal, New York
  - Luxe Vision and Optical, Powell, Ohio
  - Dr. David W. Ferris & Associates, Warwick, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu